CLINICAL TRIAL: NCT06853509
Title: Development and Validation of a Prediction Model for Predicting Gastric Neoplasia in Patients with High-risk Endoscopic Features: a Prospective Cohort Study
Brief Title: Predicting Gastric Neoplasia in Patients with High-risk Endoscopic Features
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhijun Bao, Director, Fudan University
Other Study IDs: 2024K339-F251
Record Dates: First submitted 2025-02-09; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Gastric Neoplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High-risk endoscopic features: Patients found active Helicobacter pylori infection or atrophic gastritis in initial esophagogastroduodenoscopy.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No Intervention: Observational Cohort

SUMMARY:
A prospective, single-center, cohort study to development and validation of a prediction model for predicting gastric neoplasia in patients with high-risk endoscopic features

DETAILED DESCRIPTION:
1. Patients at high risk for gastric cancer are undergone screening esophagogastroduodenoscopy at the Endoscopy department of Gastrointestinal endoscopy center of Huadong hospital affiliated to Fudan University.
2. For every enrolled patient, follow-up esophagogastroduodenoscopy were conducted in the 3rd and 5th years after the baseline examination. If high-risk endoscopic features for gastric cancer (i.e., active Helicobacter pylori infection or atrophic gastritis classified as C2-O3 according to the Kimura-Takemoto classification) were observed during the baseline examination, an additional follow-up esophagogastroduodenoscopy was performed in the 1st year after the baseline examination.
3. Clinical characteristics, gastric neoplasia-related blood biomarkers, the extent of atrophic gastritis and other endoscopic findings were collected in baseline and follow-up esophagogastroduodenoscopy. For patients whose baseline esophagogastroduodenoscopy indicates open-type atrophic gastritis (Kimura-Takemoto classification O1-O3), blood samples will be collected for whole-genome sequencing at the time of the baseline and the final follow-up examination.
4. Enrolled patients were followed up until gastric neoplasia was detected, up to a maximum of 5 years.
5. After the study was completed, a prediction model for predicting gastric neoplasia in patients with atrophic gastritis was developed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years
2. Meets the definition of a high-risk population for gastric cancer, which includes one or more of the following: (1) Residence in a high-incidence region for gastric cancer (2) Helicobacter pylori (Hp) infection (3) History of chronic atrophic gastritis, gastric ulcer, gastric polyps, post-gastrectomy status, hypertrophic gastritis, pernicious anemia, or other precancerous gastric conditions (4) First-degree relatives of patients with gastric cancer (5) Other risk factors for gastric cancer such as high salt intake, frequent consumption of pickled foods, smoking, or heavy alcohol use
3. No gastric cancer or precancerous lesions detected on initial esophagogastroduodenoscopy, yet with endoscopic features consistent with high-risk endoscopic features. High-risk endoscopic include: (1) Active Helicobacter pylori infection (2) Atrophic gastritis (Kimura-Takemoto classification C1-O3)
4. Provision of written informed consent and agreement to comply with the follow-up requirements specified in the study protocol

Exclusion Criteria:

1. Emergency esophagogastroduodenoscopy
2. History of partial or total gastrectomy
3. ASA physical status classification of 3 or higher
4. Use of oral antiplatelet or anticoagulant medications, or coagulopathy (defined as a platelet count < 50 × 10^9/L or INR > 1.5)
5. Pregnancy or lactation
6. Severe cardiac, pulmonary, hepatic, or renal disease
7. Concomitant other malignant tumors or severe infectious diseases
8. Refusal to sign the informed consent form or any other condition deemed unsuitable for study participation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with high-risk endoscopic features
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of gastric neoplasia | 2 weeks after the last follow-up
  Detection rate of gastric neoplasia during follow-up. Gastric neoplasia was defined as low-grade intraepithelial neoplasia, high-grade intraepithelial neoplasia, and adenocarcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Huadong hospital affiliated to Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after completion of this study
Access Criteria: All researchers can require the original data from principal investigator of this study (Email address: arctg4@163.com)